CLINICAL TRIAL: NCT02435732
Title: A Phase I, Single Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Tolerability of C1 Inhibitor (CINRYZE) as a Donor Pre-treatment Strategy in Brain Dead Donors Who Meet a Kidney Donor Risk Index (KDRI) Above 60%
Brief Title: CINRYZE as a Donor Pre-treatment Strategy in Kidney Recipients of KDPI>60%
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-0195; A539742 (Other: UW Madison); SMPH/SURGERY/TRANSPLANT (Other: UW Madison); Protocol Version 5/28/2018 (Other: UW Madison)
Record Dates: First submitted 2015-04-21; First posted 2015-05-06 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Heparin; SERPING1 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Standard donor management + vehicle treatment (n=9)- placebo saline solution
  Interventions: Drug: Placebo saline solution
- CINRYZE 200 U/Kg IV (Experimental): Intervention is CINRYZE 200 U/Kg IV single dose
  Interventions: Drug: Placebo saline solution; Drug: CINRYZE
- 200 units/kg IV CINRYZE with Heparin 20 U/kg/h IV (Experimental): CINRYZE 200 units/kg IV single dose with Heparin at 20 units/kg/h IV maintenance until organ recovery
  Interventions: Drug: Placebo saline solution; Drug: Heparin; Drug: CINRYZE

INTERVENTIONS:
Drug: Placebo saline solution — saline solution
Drug: Heparin — Added to the one of the arms receiving 200U/kg dose of CINRYZE
  Arms: 200 units/kg IV CINRYZE with Heparin 20 U/kg/h IV
Drug: CINRYZE — 200U/kg IV dose with or without heparin, or 500U/kg IV dose
  Other Names: C1INH
  Arms: 200 units/kg IV CINRYZE with Heparin 20 U/kg/h IV; CINRYZE 200 U/Kg IV

SUMMARY:
Limiting brain death-induced organ injury through a systemic anti- inflammatory medical management should allow for improvement in the quality of transplanted organs, and as a result, clinical improvement in post-transplant outcomes represented by a decrease in the incidence of delayed graft function (DGF) after transplantation.

The specific aim is to evaluate the effect of C1INH (CINRYZE) as a donor pre-treatment strategy to decrease systemic inflammation and decrease the incidence of DGF in Expanded Criteria Donors (ECD), currently identified as donors with Kidney Donor Profile Index (KDPI) greater than or equal to 60%.

DETAILED DESCRIPTION:
This is a randomized, single-center double-blinded study.

Donor Pre-treatment Strategy:

The main objective is to identify the lowest dose that will allow an at least 80% decrease in the activity of classic pathway and Mannose-Binding Lectin (MBL) pathway of complement. The main objectives parallel observations in non-human primates in which animals receiving kidneys from donors in which activity of both classic and MBL pathways of complement were reduced by at least 50% with the use of C1 inhibitors displayed very mild or no delayed graft function after transplantation.

This trial has specifically been designed to evaluate the beneficial effect of C1INH in kidneys from deceased donors which have a high rate of delayed graft function. The selection of potential donors to be part of this study will be limited to the population of donors with a KDPI over 60%.

A total of 36 brain dead donors and 72 kidney recipients will be included in the study.

Most of the donors with a Kidney Donor Profile Index (KDPI) >60%, due to the fact that they are considered "extreme" donors, are not likely to be able to donate organs other than kidneys. They would certainly not be pancreas donors, and it is unlikely they would be lung donors. There is a small possibility that donors with a KDPI >60% could be potential liver donors. In the event that a donor liver is available for transplant, we will obtain written consent from the liver recipient, as we will from the kidney recipient(s) before the donor is dosed with the CINRYZE/placebo.

For this study:

All donors will come from within our service area. All kidney and livers will be allocated to be transplanted at the UW.

Stage 1: Collection of initial safety data prior to expanding the study to a broad cohort of patients.

3 non-randomized donors: Step 1: Two kidney only donors treated with 200 units/kg C1INH and heparin at 20 units/kg/h IV maintenance until organ recovery Step 2: Two donors of both liver and kidneys, treated with 200 units/kg C1INH and heparin at 20 units/kg/h IV maintenance until organ recovery The 8 kidneys and 2 livers in Stage 1 will be allocated to be transplanted only at UW.

Stage 2: PK Study, Safety and Outcome Data

36 donors will be randomized into 3 groups:

Group 1: Control group: standard donor management + vehicle treatment (n=12) Group 2: Standard donor management + C1INH at a dose of 200 U/Kg IV single dose (n=12) Group 3: Standard donor management + C1INH at a dose of 200 units/kg IV single dose and heparin at 20 units/kg/h IV maintenance until organ recovery (n=12)

ELIGIBILITY:
Inclusion Criteria for Kidney Recipient:

* Adult patients receiving a kidney from a donor with KDPI>60%
* Provide written informed consent.
* Accepted for renal transplantation due to end stage renal disease (Chronic Kidney Disease Stage V).
* Recipient of a first or second renal transplant.
* For second renal transplantation, minimum 3 months since the loss of the first transplanted kidney.
* At least 18 years of age:

If female, patient must be/have:

* Post-menopausal, defined as the absence of menses for at least one year (serum FSH ≥20I U/L can also be measured according to local practice), OR Surgically sterile, defined as a bilateral tubal ligation at least 6 months prior to administration of study drug, bilateral oophorectomy, or complete hysterectomy, OR Using an effective means of contraception (per Appendix 1) that is planned to continue for the duration of the study (one year), AND negative urine pregnancy test if the patient is capable of providing a urine sample. If not capable to provide urine sample, serological pregnancy test will be perform.
* Female patients of childbearing potential who are anuric must have a serum pregnancy test.

If male, patient must:

* Agree to use an effective means of contraception (per site-specific guidelines) that is planned to continue for the duration of the study (6 months).
* Agree not to donate sperm until 6 months after dosing.

Patients must be willing to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations.

Inclusion Criteria for Liver Recipients*:

* Provide written informed consent.
* Accepted for liver transplantation
* Recipient of a first liver transplant.
* At least 18 years of age:

If female, patient must be/have:

* Post-menopausal, defined as the absence of menses for at least one year (serum FSH ≥20I U/L can also be measured according to local practice), OR
* Surgically sterile, defined as a bilateral tubal ligation at least 6 months prior to administration of study drug, bilateral oophorectomy, or complete hysterectomy, OR
* Using an effective means of contraception (per Appendix 1) that is planned to continue for the duration of the study (one year), AND negative urine pregnancy test if the patient is capable of providing a urine sample. If not capable to provide urine sample, serological pregnancy test will be perform.
* Female patients of childbearing potential who are anuric must have a serum pregnancy test.

If male, patient must:

* Agree to use an effective means of contraception (per site-specific guidelines) that is planned to continue for the duration of the study (one year).
* Agree not to donate sperm until 6 months after dosing.

  * Willingness to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations.

The criteria for enrollment in the study was originally limited to kidney donors with KDPI >85%. Over the last five years however, we have only transplanted a handful of those patients If we further restrict our patient pool to those who are not liver donors, our pool of possible donors will become even smaller, making the study very difficult, if not impossible, to complete. Furthermore, our knowledge of the pathophysiology of the complement system suggests that use of C1Inhibitor will improve liver outcomes by blunting the inflammatory response which can cause liver fibrosis and reperfusion injury. Since we have seen no negative effects on the liver in our preliminary non-human primate data, there is no need to exclude possible liver donors from our treatment.

Therefore, in order to increase feasibility of the study, we have now expanded the trial to include donors with a KDPI above 60% (rather than > 85%), since the rate of DGF in recipients of kidneys from KDPI between 60% and 85% is similar to the group >85%. In addition, we are now including liver recipients in the study, and will consent them if the donor has a viable liver in addition to the kidney(s). If we were to only include patients with KDPI above 85%, and kidney only donors, this trial would not be feasible.

Exclusion Criteria:

* Use of an investigational drug in the 30 days before surgery.
* Participation in any other research study (drug or non-drug) without prior approval from the Medical Monitor.
* Known hypersensitivity to human monoclonal antibodies or any of the study drug excipients.
* Previous hypersensitivity to basiliximab, Campath-1H or antithymocyte globulin (ATG)
* History of or known HIV, HBV (surface antigen), or HCV positivity
* History of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin, or cervical intraepithelial neoplasia.
* Scheduled to undergo multi-organ transplantation.
* Presence of clinically significant infections requiring continued therapy.
* Positive screening for active tuberculosis.
* Existence of any surgical or medical condition, other than the current transplantation which, in the opinion of the investigator, might significantly alter the distribution, metabolism or excretion of study medication.
* History or presence of a medical condition or disease that in the investigator's assessment would place the patient at an unacceptable risk for study participation.
* Lactating or pregnant woman.
* Patient institutionalized by administrative or court order.
* HLA or ABO incompatible kidney defined as a positive cytotoxic crossmatch, positive mean fluorescent intensity beyond the acceptable parameters by the institution, or flow crossmatch-based assay that is positive (for kidney recipients only)

Exclusion Criteria for Brain Dead Donor:

* Donor who is known to have received an investigational drug for I-R injury or graft rejection (immunosuppressant) in the 48H prior to organ recovery
* Participation in any other research study (drug or non-drug) without prior approval from the PI
* Donor institutionalized by administrative or court order
* Donors whose organs are allocated for transplantation to other transplant programs outside UW
* Donors for which any of the intended organ recipients has not provided consent for the study
* Donors that are donating other organs outside the scope of the study (i.e. heart, lungs, intestine) will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Lowest dose that will allow at least an 80% decrease in the activity of classic pathway and MBL pathway of complement in brain death donors with KDPI over 60%, with the purpose of reducing the incidence of delayed graft function. | over a 12 month period
  Assessment of graft function

SECONDARY OUTCOMES:
Donor Pharmacokinetics: plasma concentrations and Area under the Curve (AUC) for CINRYZE | At various timepoints within first 24 hours
  pharmacokinetics
Rate of of DGF in kidney transplantation from ECD brain death donors | Within 6 hours of brain death
  DGF rate
Level of suppression of the classical and MBL pathways | Within 6 hours of brain death
  classical and MBL pathways
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day of Transplant: first 24 hours, days 2-7, weeks 2,3,8, month 3, 6, 12
  Safety and tolerability
Levels of complement activation after brain death in donors treated with C1INH | Within 6 hours of brain death
  Complement activation

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fernandez, MD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No